CLINICAL TRIAL: NCT05941403
Title: Developing and Testing a Produce Prescription Implementation Blueprint to Improve Food Security in a Clinical Setting: A Pilot Study
Brief Title: Developing and Testing a Produce Prescription Implementation Blueprint to Improve Food Security in a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Peter G. Peterson Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000018; 008225 (Other Grant/Funding Number: Peter G. Peterson Foundation)
Record Dates: First submitted 2023-06-09; First posted 2023-07-12 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Food Insecurity
Keywords: food insecurity; implementation science; produce prescription program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced Produce Prescription Implementation (Experimental): The study team will develop an enhanced implementation blueprint to support uptake of the produce prescription (VeggieRx) intervention that is informed by advisory board input and includes multiple implementation strategies to address identified barriers to implementation.
  Interventions: Behavioral: Enhanced Produce Prescription Implementation

INTERVENTIONS:
Behavioral: Enhanced Produce Prescription Implementation — Practices make modifications to their usual produce prescription program based on an implementation blueprint. While the exact implementation strategies to be added will be defined based on qualitative data (data collection in progress), possible implementation strategies may include training or technical assistance.

SUMMARY:
The goal of this pilot feasibility implementation trial is to assess preliminary feasibility and acceptability of a set of produce prescription implementation strategies. Produce prescription programs are one approach to addressing food insecurity, or the lack of adequate access to safe and nutritious foods. Produce prescriptions involve healthcare providers identifying patients at risk for food insecurity and writing prescriptions for those patients to receive subsidized vegetables. In this study, the investigators will work with a community advisory board to develop a set of enhanced implementation strategies (e.g., training, technical assistance) to support healthcare providers in delivering produce prescription programs. The investigators will assess the feasibility, acceptability, and appropriateness of these strategies. Pre-post changes in implementation outcomes (i.e., adoption) and effectiveness outcomes (i.e., food security) will be examined.

DETAILED DESCRIPTION:
Healthcare providers/staff and patients will be recruited from allied Integra health centers. Following enrollment in the already existing produce prescription program ("VeggieRx"), participants will be asked if they would be interested in participating in the research study that entails surveys regarding the program. The investigators expect to recruit participants into the study starting shortly after patients get enrolled in the program. Potential participants will be informed that their decision about whether to participate in the research study will not affect their eligibility or enrollment in the VeggieRx program. They will also be informed that this study seeks to understand strategies to improve the current VeggieRx program. A research assistant will follow-up with interested patients/providers/staff and complete enrollment, consents, and a baseline assessment, either in the waiting room to complete on their own, over the phone or Zoom, OR if they choose to complete it on their own, the study team will send them the link to the consent and survey. It should be noted that participants can either choose to complete the surveys on their own through a survey link (which will be the default) or the surveys can be administered by the study staff. The study team hopes to collect baseline measures before the delivery of their first vegetables which typically begins the second week in July. While providers/staff will not be receiving vegetables, the study team also hopes to collect their baseline data when the program begins (by second week of July). Follow-up data collection for patients will occur after their final delivery (usually end of November) and provider/staff survey will also occur around that time. The study team will communicate with the program to find out when the last deliveries are occurring (not gathering any patient information, just overall timeline).

Baseline and final measures for participating patients are each expected to take approximately 15-20 minutes. In addition, VeggieRx participants will also complete a biweekly measure of engagement which will take approximately 2-minutes each time and will be sent via text message or email depending on participants' preferences throughout the duration of the 6-month VeggieRx delivery period. These questions will ask if they received their vegetable delivery, how much they liked the vegetables, how much they used them and if they fit with their families' eating habits.

As described above, providers and staff will be contacted via email/text/phone by the research assistant asking them to participate. They can complete measures with a research assistant or on their own. Baseline and follow-up surveys for providers/staff are each expected to take 10-20 min. All previously mentioned study procedures can take place in Spanish for patients whose primary language is Spanish by the research assistant research staff that is fluent in Spanish.

ELIGIBILITY:
Healthcare providers/staff Inclusion Criteria:

* 18 years of age or older
* healthcare provider/staff member who makes referrals to produce prescriptions (VeggieRx)
* fluent in English and/or Spanish

Healthcare providers/staff Exclusion Criteria

* under age 18
* have not been involved in referral process for produce prescriptions (VeggieRx)
* are not fluent in English and/or Spanish

Patient Inclusion Criteria:

* 18 years of age or older
* enrolled in the produce prescription program (VeggieRx)
* fluent in English and/or Spanish

Patient Exclusion Criteria:

* under age 18
* declined to enroll in the produce prescription program (VeggieRx)
* are not fluent in English and/or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Engagement with the Produce Prescription Program Questionnaire | Baseline
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores on each item indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 2
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 4
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 6
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 8
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 10
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 12
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 14
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 16
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 18
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 20
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 22
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 24
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 26
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Patient Engagement with the Produce Prescription Program Questionnaire | Week 28
  Patient engagement will be measured with a 4-question biweekly questionnaire that includes items rated on a 5-point (1-5) Likert-scale related to whether patients received the produce and whether they used it and liked it. Higher scores indicate higher engagement. Scores range from 4-20.
Acceptability of Intervention Measure | Baseline
  Acceptability of produce prescriptions will be assessed using the 4-item Acceptability of Intervention measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Higher scores indicate higher acceptability of the intervention. Scores range from 4-20.
Acceptability of Intervention Measure | 6 month follow up
  Acceptability of produce prescriptions will be assessed using the 4-item Acceptability of Intervention measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Higher scores indicate higher acceptability of the intervention. Scores range from 4-20.
Feasibility of Intervention Measure | Baseline
  Feasibility of produce prescriptions will be assessed using the 4-item Feasibility of Intervention Measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Higher scores indicate higher feasibility of the intervention. Scores range from 4-20.
Feasibility of Intervention Measure | 6 month follow up
  Feasibility of produce prescriptions will be assessed using the 4-item Feasibility of Intervention Measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Higher scores indicate higher feasibility of the intervention. Scores range from 4-20.
Intervention Appropriateness Measure | Baseline
  Appropriateness of produce prescriptions will be assessed using the 4-item Intervention Appropriateness Measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Higher scores indicate higher appropriateness of the intervention. Scores range from 4-20.
Intervention Appropriateness Measure | 6 month follow up
  Appropriateness of produce prescriptions will be assessed using the 4-item Intervention Appropriateness Measure with scores ranging from 1 (completely disagree) to 5 (completely agree). Higher scores indicate higher appropriateness of the intervention. Scores range from 4-20.
Evidence-Based Practice Attitudes Scale | 6-month follow up
  The Evidence-Based Practice Attitudes Scale measures providers' attitudes toward evidence-based practices - specifically produce prescription programs. Scores range from 0 (not at all) to 4 (to a very great extent); higher scores indicate more positive attitudes toward evidence-based practices. Scores are calculated as an average and range from 0-4.
Feasibility of Participant Enrollment | Baseline
  Proportion of participants who agree to enroll in the study out of those who are enrolled in the produce prescription program
Implementation Climate Scale | 6 month follow up
  This measure of implementation climate will assess the innovation-specific organizational climate for implementing produce prescription programs. Responses will be rated on a 4-point scale ranging from 0 (not at all) to 4 (very great extent). Higher responses indicate a stronger implementation climate. Scores are calculated as an average and range from 0-4.
Implementation Readiness: Organizational Readiness for Implementing Change | Baseline
  This measure will assess organizations' readiness to implement a new intervention. Responses will be rated on a 5 point scale ranging from 1 (disagree) to 5 (agree). Higher scores indicate higher organizational readiness for change. Scores range from 12-60.
Implementation Readiness: Organizational Readiness for Implementing Change | 6-month follow up
  This measure will assess organizations' readiness to implement a new intervention. Responses will be rated on a 5 point scale ranging from 1 (disagree) to 5 (agree). Higher scores indicate higher organizational readiness for change. Scores range from 12-60.

SECONDARY OUTCOMES:
Adoption of Produce Prescriptions | Baseline
  Number of patients who enroll in the produce prescription program
Adoption of Produce Prescriptions | 6 month follow up
  Number of patients who enroll in the produce prescription program
Effectiveness: Food Security | Baseline; 6 month follow up
  Measured by the 6-item United States Department of Agriculture measure. Total scores range from 0-6, with lower scores indicating food security.
Effectiveness: Food Security | Baseline
  Measured by the 6-item United States Department of Agriculture measure. Total scores range from 0-6, with lower scores indicating more food security.
Effectiveness: Nutrition security | 6 month follow up
  measured by the 4-item Nutrition Security measure. Responses range from "never" (0) to "always" (4). Items are scored by finding a mean of included items. Lower scores indicate more nutrition security.
Effectiveness: Patient Health Questionnaire-2 | baseline, 6-month follow up
  The 2-item Patient Health Questionnaire will be used to screen for depression. Responses range from 0 (not at all) to 3 (nearly every day). Scores greater than 3 suggest that major depressive disorder is likely.
Effectiveness: Patient Health Questionnaire-2 | 6-month follow up
  The 2-item Patient Health Questionnaire will be used to screen for depression. Responses range from 0 (not at all) to 3 (nearly every day). Scores greater than 3 suggest that major depressive disorder is likely.
Effectiveness: Dietary Screener Guide | baseline, 6-month follow up
  Fruit and vegetable intake will be measured by the 10-item Dietary Screener Guide, in which participants will be asked to rate the frequency with which they have eaten a variety of foods. Responses range from "never" to "6 or more times per day." The measure is scored using a scoring algorithm that converts survey responses to estimates of average daily dietary intake for fruits and/or vegetables.
Effectiveness: Dietary Screener Guide | 6-month follow up
  Fruit and vegetable intake will be measured by the 10-item Dietary Screener Guide, in which participants will be asked to rate the frequency with which they have eaten a variety of foods. Responses range from "never" to "6 or more times per day." The measure is scored using a scoring algorithm that converts survey responses to estimates of average daily dietary intake for fruits and/or vegetables.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah E Frank, PhD, Principal Investigator — Brown University; Alison Tovar, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Brown Research on Implementation and Dissemination to Guide Evidence use (BRIDGE) Program, Providence, Rhode Island
  - Department of Behavioral and Social Sciences/School of Public Health, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
Given the small dataset, data will not be made publicly available. However, de-identified quantitative data will be made available to individual investigators following a written request to the study principal investigators.

REFERENCES:
- [Background] Frank HE, Guzman LE, Ayalasomayajula S, Albanese A, Dunklee B, Harvey M, Bouchard K, Vadiveloo M, Yaroch AL, Scott K, Tovar A. Developing and testing a produce prescription implementation blueprint to improve food security in a clinical setting: a pilot study protocol. Pilot Feasibility Stud. 2024 Mar 23;10(1):51. doi: 10.1186/s40814-024-01467-7. PMID 38521931

DOCUMENTS (1):
  • Informed Consent Form (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT05941403/ICF_000.pdf